CLINICAL TRIAL: NCT03439540
Title: The Study on the Influence of Plantago Species (Plantago Major) on Adipose Tissue Content, Mineral Metabolism and Other Selected Biochemical Parameters of Blood in Obese Women
Brief Title: Influence of Plantago Major on Mineral Metabolism and Selected Biochemical Parameters in Obese Women
Acronym: Plantago
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Joanna Suliburska, assiastant professor, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1104/16
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Obesity
Keywords: Plantago major; obesity; mineral content; adipose tissue
MeSH Terms: conditions — Obesity | interventions — sucrose transport protein, plant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Individuals receive a placebo daily, for 12 weeks.
  Interventions: Dietary Supplement: Placebo
- Plantago major (Experimental): Individuals receive Plantago major daily, for 12 weeks.
  Interventions: Dietary Supplement: Plantago major

INTERVENTIONS:
Dietary Supplement: Plantago major — Individuals receive Plantago major daily, for 12 weeks
  Arms: Plantago major
Dietary Supplement: Placebo — Individuals receive placebo daily, for 12 weeks
  Arms: Placebo

SUMMARY:
Effect of oral supplementation with Plantago major on cardiometabolic risk factors and mineral content and lifestyle in obese women: double-blind, randomized clinical trial.

DETAILED DESCRIPTION:
The purpose of the study is to determine whether oral Plantago major supplementation affects cardiometabolic risk factors, mineral content, and lifestyle in obese women.

In previous research it was found that the Plantago maxima extract counteracts the development of adipose tissue in rats on a high-fat diet. In addition, antioxidative, anti-inflammatory and antidiabetic action of Plantago has been demonstrated. Moreover, it has been shown that Plantago influences lipolysis in obese mice and ameliorates metabolic processess in obese rats.

The project is due to evaluate the effect of oral supplementation with selected Plantago species - Plantago major in obese patients on:

* the content of minerals in blood, hair and urine
* total cholesterol, HDL and LDL cholesterol and triglycerides blood concentration,
* blood glucose and insulin concentration,
* blood pressure,
* anthropometric parameters: body mass, body height, waist and hip circumferences
* body content measured by bioimpedance: % of fat tissue and % of muscle tissue
* quality of life

  70 subjects will be randomized into two groups and receive oral Plantago major extract (the first group) or oral placebo (the second group) once daily for 12 weeks. At baseline and at completion (after 12 weeks) fasting blood, urine and hair samples will be collected and abovementioned parameters will be measured.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) equal to or greater than 30 kg/m2

  * age 18 to 60 years
  * stable body weight (< 3 kg self-reported change during the previous three months)
  * written informed consent to participate in the study,
  * abdominal obesity - waist circumference> 80 cm;
  * body fat content measured by bio-impedance ≥ 33%;
  * female

Exclusion Criteria:

* secondary obesity or secondary hypertension
* diabetes type I
* gastrointestinal disease;
* dyslipidaemia, type 2 diabetes, hypertension requiring the implementation of pharmacological treatment in the last 3 months prior to observation or follow-up;
* a history of use of any dietary supplements within the one month prior to the study
* clinically significant acute or chronic inflammatory disease in the respiratory, gastrointestinal or genitourinary system or in the mouth, throat, paranasal sinuses and / or connective tissue disease, arthritis;
* simultaneous participation in a study that affects body mass or use of diet / medication / nutritional behaviors affecting body mass;
* a history of infection in the month prior to the study
* nicotine, drug or alcohol abuse
* or other condition that, in the opinion of the investigators, would make participation not in the best interest of the patient or could prevent, limit, or confound the study results

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
mineral content | At the baseline and following 12 weeks of treatment
  content of minerals in serum, urine and hair

SECONDARY OUTCOMES:
blood pressure | At the baseline and following 12 weeks of treatment
  blood pressure
body mass | At the baseline and following 12 weeks of treatment
  body mass
body height | At the baseline and following 12 weeks of treatment
  body height
hip circumference | At the baseline and following 12 weeks of treatment
  hip circumference
waist circumference | At the baseline and following 12 weeks of treatment
  waist circumference
body content measured by bioimpedance: % of fat tissue | At the baseline and following 12 weeks of treatment
  Content of fat tissue measured by bioimpedance
body content measured by bioimpedance: % of muscle tissue | At the baseline and following 12 weeks of treatment
  Content of muscle tissue measured by bioimpedance
serum total cholesterol | At the baseline and following 12 weeks of treatment
  Serum concentration of total cholesterol
serum LDL cholesterol | At the baseline and following 12 weeks of treatment
  Serum concentration of LDL cholesterol
serum HDL cholesterol | At the baseline and following 12 weeks of treatment
  Serum concentration of HDL cholesterol
serum triglycerides | At the baseline and following 12 weeks of treatment
  Serum concentration of triglycerides
insulin | At the baseline and following 12 weeks of treatment
  insulin serum concentration
glucose | At the baseline and following 12 weeks of treatment
  glucose serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Suliburska, Assoc. Prof., Principal Investigator — Poznan University of Life Sciences
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland